CLINICAL TRIAL: NCT00721201
Title: A Pilot Study of the Effect of a Glucocorticoid Receptor Antagonist in Patients With Subclinical Cushings
Brief Title: Glucocorticoid Receptor Antagonism in Subclinical Cushings
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: HRA Pharma (Industry)
Responsible Party: Dr John Newell-Price, University of Sheffield
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH14791
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Subclinical Cushing's
Keywords: subclinical Cushing's
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mifepristone — Use of mifepristone 200mg bd for 8 weeks

SUMMARY:
The purpose of this study is to assess the effects of reducing the activity of endogenous glucocorticoid in patients with low-grade cortisol excess

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion if: they are males and over 18, lack clinical features classically associated with Cushing's syndrome; have evidence of excess circulating cortisol

Exclusion Criteria:

* Evidence of local or systemic malignancy; overt Cushing's syndrome; severe uncontrolled diabetes mellitus or hypertension; pregnancy; clinically significantly impaired cardiovascular function (e.g. stage IV cardiac failure); severe liver disease (liver enzymes ≥ 3 x the institutional upper limit of normal range); significantly impaired renal function (eGFR <30/min); uncontrolled severe active infection; treatment with approved or experimental steroidogenesis inhibitors, adrenolytic agents, within four weeks of admission; In women, known endometrial cancer, history of endometrial hyperplasia or vaginal bleeding of unknown cause; requirement for inhaled or systemic glucocorticoids for existing disease; impaired mental capacity or markedly abnormal psychiatric evaluation that precludes informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks

SECONDARY OUTCOMES:
Glucose homeostasis | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr John Newell Price, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

REFERENCES:
- [Derived] Debono M, Chadarevian R, Eastell R, Ross RJ, Newell-Price J. Mifepristone reduces insulin resistance in patient volunteers with adrenal incidentalomas that secrete low levels of cortisol: a pilot study. PLoS One. 2013;8(4):e60984. doi: 10.1371/journal.pone.0060984. Epub 2013 Apr 5. PMID 23577182